CLINICAL TRIAL: NCT06462950
Title: Study 3: The Experimental Examination of Ostracism and Concealability on Gendered Stigma Smoking Outcomes
Brief Title: Experiment Among Smokers in Which Two Variables Are Manipulated: Ostracism and Concealability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dickinson College (Other)
Responsible Party: Principal Investigator, Marie Helweg-Larsen, Professor, Dickinson College
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: MHLStudy3
Record Dates: First submitted 2024-06-04; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Ostracism
Keywords: stigmatization
MeSH Terms: conditions — Ostracism; Stereotyping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ostracism (Experimental): Ostracism is manipulated by randomly assigning people to the inclusion condition (they play an online ball tossing game and get the ball passed a third of the time) or exclusion condition (they get the ball passed twice in the beginning of the game and then not again).
  Interventions: Behavioral: Do men and women differ in their reactions to the experimental conditions.
- Concealment (Experimental): Concealment is manipulated by randomly assigning the participants to information that the other players did (revealed condition) or did not know (concealed condition) the gender of the participant.
  Interventions: Behavioral: Do men and women differ in their reactions to the experimental conditions.

INTERVENTIONS:
Behavioral: Do men and women differ in their reactions to the experimental conditions. — Do men and women differ in their reactions to the experimental conditions.

SUMMARY:
The goal of this experimental study is to learn about the effects of ostracism and concealment among adult smokers. The main aims are:

1. Determine the causal consequences of gendered stigmatization. Specifically, do women react more strongly than men to exclusion (as opposed to inclusion) especially when their gender is revealed (as opposed to concealed) for outcomes such as smoking stigma, stress, cognitive depletion, smoking attitudes, and smoking cessation intentions (Study 3)?
2. Examine the moderating roles of cultural context. Specifically, contrasting the cultural context in the US and Denmark (where gender norms are more egalitarian) do Danish smokers show fewer gender differences than US smokers in how they describe and react to their smoking stigmatization experiences (Study 1, 2, and 3)?

DETAILED DESCRIPTION:
The proposed studies examine cross-culturally the reasons why among smokers, women feel more stigmatized than men do. An experiment with US and Danish smokers will examine how men and women differ in their reactions to being stigmatized (using a standard exclusion manipulation) when their gender is revealed instead of concealed. The outcome measures will include stress, smoking stigma, cognitive depletion, smoking attitudes, and smoking cessation intentions.

ELIGIBILITY:
Inclusion Criteria:

* daily smoker who smoker more than 5 cigarettes daily and have smoked for at least 1 year
* speak English reside in the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation of gender identit
Enrollment: 340 (Estimated)
Dates: Start 2028-05 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive depletion | 10 min
  The Stroop Color-Word Interference Test measures the executive control needed to suppress reading a word and instead naming the color of the word. The test will be adminstered once immediately after the experimental task.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code